CLINICAL TRIAL: NCT06626035
Title: Prospective Randomized Evaluation of Analgesia for Cardiac Elective Surgery in Children (PRECISE Cardiac Trial)
Brief Title: Evaluation of Analgesia for Cardiac Elective Surgery in Children
Acronym: PRECISE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Senthil Sadhasivam (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24040108; U01HD116257 (NIH)
Record Dates: First submitted 2024-06-15; First posted 2024-10-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cardiac Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methadone-Based ERAS Group (Experimental): The methadone-based standardized analgesia intervention arm will include standardized perioperative care and analgesia, including intraoperative intravenous methadone (1st dose: 0.1 mg/kg up to a maximum of 5 mg before incision; 2nd dose: 0.1 mg/kg up to a maximum of 5 mg 4 hours after 1st dose) and postoperatively, up to 4 oral or IV doses of methadone (0.1 mg/kg up to a maximum of 5 mg) every 12 hours before discharge as part of standardized multimodal analgesia in the hospital setting.
  Interventions: Drug: Methadone based ERAS
- Non-Methadone-Based Group (Active Comparator): Children randomized to the standard-of-care arm will receive standard opioid analgesia protocol without intra- and post-operative methadone per the current site standards.
  Interventions: Drug: Non-methadone based group

INTERVENTIONS:
Drug: Methadone based ERAS — Children randomized to the methadone arm will include standardized perioperative care and analgesia, including intraoperative intravenous methadone (1st dose: 0.1 mg/kg up to a maximum of 5 mg before incision; 2nd dose: 0.1 mg/kg up to a maximum of 5 mg 4 hours after 1st dose) and postoperatively, up to 4 oral or IV doses of methadone (0.1 mg/kg up to a maximum of 5 mg) every 12 hours before discharge as part of standardized multimodal analgesia in the hospital setting.
  Other Names: Methadone-Based
  Arms: Methadone-Based ERAS Group
Drug: Non-methadone based group — Children randomized to the standard-of-care arm will receive standard opioid analgesia protocol without intra- and post-operative methadone per the current site standards.
  Other Names: Standard Care
  Arms: Non-Methadone-Based Group

SUMMARY:
The purpose of this study is to look at a standardized methadone-based enhanced recovery after surgery protocol following pediatric cardiac surgery. This study will consist of randomly assigning children to receive the methadone-based recovery procedures or to receive current standard of care recovery procedures. Randomly assigning means that there is a 50/50 chance, like a coin flip, of being assigned to either research group.

DETAILED DESCRIPTION:
Specific Aims Aim 1. Conduct a randomized clinical trial in cardiac surgery (CS) to compare acute pain relief, opioid-sparing efficacy, and safety of standardized perioperative multidose methadone-based enhanced recovery after surgery (ERAS) vs. standard-of-care non-methadone-based analgesia.

Aim 2. Develop precision methadone dosing based on age, CYP2B6 and ORM1 variants, and alpha acid glycoprotein (AAG) levels, cardio-pulmonary bypass (CPB) related dilution.

Aim 3. Identify patient profiles that predict benefits from the assigned analgesia protocol to optimize clinical outcomes. Personalized risk prediction models will be developed and validated including genetic variants (i.e., CYP2B6, CYP2D6, ABCB1, OPRM1, and FAAH), and psychological and clinical factors to predict benefit with the assigned treatments (methadone or non-methadone) for pre-specified clinical endpoints (i.e., lower acute surgical pain, respiratory depression [RD], postoperative nausea and vomiting [PONV], opioid dependence [OD], and chronic postsurgical pain [CPSP]) in cardiac surgery.

Overall Impact Investigators will develop actionable evidence for the efficacy of standardized, multidose, methadone-based ERAS protocols and will harness genetic, clinical, and psychological factors contributing to variability in methadone and oxycodone PK, acute surgical pain, transition to CPSP, opioid-induced PONV, RD, and dependence to develop personalized analgesia strategy and dosing for children undergoing cardiac surgery. Implementation of evidence-based standardized methadone-based ERAS pain management and individualized risk prediction will maximize acute surgical pain relief while minimizing opioid use and AEs in millions of children.

Hypothesis The central hypothesis is that a standardized, multidose, methadone-based ERAS protocol will reduce acute surgical pain, overall opioid use, RD, PONV and CPSP compared with standard-of-care short-acting opioid-based analgesia in children undergoing cardiac surgery. The long-term goal is to proactively improve the safety and efficacy of surgical pain control while reducing opioid AEs and the opioid epidemic burden in all children undergoing inpatient surgeries. Further, we hypothesize that age, CYP2B6 and ORM1 variants, AAG levels, and CPB-related dilution will explain methadone's PK variability and dose adjustments that correlate with optimal clinical outcomes, and that patient profiles based on genetic, psychological, and that clinical factors will predict benefits from the assigned analgesia protocol to optimize clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-years - <18 years
* ASA physical status 1, 2, or 3
* Participant or legal guardian can speak and read English or Spanish
* Undergoing the following cardiac surgeries (Categories 1 & 2) that are associated with significant acute surgical pain

STS Category 1:

* ASD, PFO closure
* VSD repairs,
* Aortic stenosis sub-valvular repair
* ASD and Partial anomalous venous return repair
* AV canal transitional
* Conduit replacement
* Valve replacement (AVR, PVR)
* TOF repair without ventriculostomy

STS Category 2:

* Glenn shunt (on Bypass only)
* Fontan surgery (on Bypass only)
* Pulmonary artery plasty (main)
* Left Atrium (LA) to Pulmonary Artery (PA) conduit replacement.

Exclusion Criteria:

* Pregnant patients
* Methadone allergy
* Preoperative prolonged QTc more than 460 msec (-30 days to 0 day)
* Subjects undergoing concomitant treatment with known cytochrome P450 inhibitors included in methadone labeling (i.e. macrolides (e.g. erythromycin), azole-antifungal agents (e.g. ketoconazole, voriconazole), protease inhibitors (e.g. ritonavir), fluconazole, SSRIs (e.g. sertraline, fluvoxamine)
* Preoperative opioid use within 30 days before surgery
* History of severe sleep apnea (have a sleep study with an AHI index score more than 10 or clinical signs of sleep disordered breathing - snoring, daytime drowsiness)
* Significant liver, kidney, neurological disease, developmental delay, or any other co-existing medical condition per discretion of the clinical investigator

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Average postoperative pain scores | Postoperative 48 hours
  Average postoperative pain scores within 48 hours of surgery (Numerical Rating Scale [NRS], or Facial expression, Leg movement, Activity, Cry, and Consolability [FLACC], both 0-10). Outcome will be reported based on area under the curve (AUC) as mean(SD).
Total postoperative opioid use | Postoperative 48 hours
  Total Opioid use in Morphine Milligram Equivalents (MME) (mg), will be reported as mean (SD).

SECONDARY OUTCOMES:
Incidence of Inpatient Respiratory Depression (RD) | Postoperative 120-hours
  RD is defined as respiratory rate <8 breaths per minute requiring oxygen in the absence of airway obstruction. Outcome measure will be reported as n(%).
Incidence of Inpatient Postoperative Nausea and Vomiting (PONV) | Postoperative 120-hours
  PONV will be assessed by self-report, EMR, and medication use. Outcome measure will be reported as n(%).
Incidence of Inpatient Sedation | Postoperative 120-hours
  Sedation will be assessed using the Ramsay Sedation Scale (RSS) and validated sedation scales extracted from the EMR. Outcome measure will be reported as n(%)
QTc Prolongation | Postoperative 48-hours
  QTc prolongation is defined as more than 460 msec. Outcome measure will be reported as n(%).
Length of Hospital Stay (LOS) | Up to 30 days
  LOS will be recorded in days. Outcome measure will be reported as mean(SD).
Persistent Opioid Use | 1-week, 1-month, and 3-months post-surgery
  Based on Prescription Drug Monitoring Program (PDMP) and self-report data. Outcome measure will be reported as n(%)
Presence of Chronic Postsurgical Pain (CPSP) at 3-months | 3-months post-surgery
  CPSP incidence will be defined using NRS pain >3/10 and functional limitations based on Functional Disability Inventory (FDI). NRS pain scores are on a scale of 0=no pain at all and 10=worst pain imaginable. Outcome measure will be reported as n(%)
Presence of Opioid Dependence (OD) at 3-months | 3-months post-surgery
  OD will be assessed using PROMIS and Prescription Pain Medication Misuse (PPMM). Outcome measure will be reported as n(%).

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiable data and specimens will be shared with the sponsor of the study. The investigators and the study team will comply with all the NIH's Public Access and Data Sharing requirements including Release of Publications and Sharing of Underlying Primary Data. Release of Publications: The investigators will publish their results in open access journals for broad and free availability immediately without any embargo period. Electronic copies of publications will be deposited within four weeks of acceptance by a journal in PubMed Central with proper metadata to be made discoverable and accessible upon publication.
Supporting Information: Study Protocol, SAP
Time Frame: Time frame is within 5-years of study completion.
Access Criteria: Online collaborative tools to facilitate data sharing such as SharePoint or Xythos